CLINICAL TRIAL: NCT04812730
Title: Multimodal Bio-mechanical Analysis of Adult Spinal Deformity With Sagittal Plane Misalignment
Acronym: ASD
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Universitaire Ziekenhuizen KU Leuven (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: S58082
Record Dates: First submitted 2021-03-18; First posted 2021-03-24 (Actual); Last update posted 2024-11-08 (Actual); Status verified 2024-11

CONDITIONS: Spinal Deformity
Keywords: Sagittal plane misalignment; Trunk and lower limb; Motion analysis; EOS stereo radiography

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- ASD with decompensated sagittal misalignment (Other): Adults suffering from a spinal deformity with a decompensated sagittal misalignment
  Interventions: Other: 2D versus 3D analysis of EOS stereo radiographic analysis; Other: Static versus dynamic analysis; Other: Pre- versus postoperative analysis; Other: Reliability of the dynamic evaluation
- ASD with compensated sagittal misalignment (Other): Adults suffering from a spinal deformity with a compensated sagittal misalignment
  Interventions: Other: 2D versus 3D analysis of EOS stereo radiographic analysis; Other: Static versus dynamic analysis; Other: Pre- versus postoperative analysis; Other: Reliability of the dynamic evaluation
- ASD without sagittal misalignment (Other): Adults suffering from a spinal deformity without a sagittal misalignment
  Interventions: Other: 2D versus 3D analysis of EOS stereo radiographic analysis; Other: Static versus dynamic analysis; Other: Pre- versus postoperative analysis; Other: Reliability of the dynamic evaluation
- Control group (Other): Asymptomatic adults not suffering from a spinal deformity
  Interventions: Other: 2D versus 3D analysis of EOS stereo radiographic analysis; Other: Static versus dynamic analysis; Other: Reliability of the dynamic evaluation

INTERVENTIONS:
Other: 2D versus 3D analysis of EOS stereo radiographic analysis — The use of EOS stereo radiographic analysis and health related quality of life scores to measure the distance of the center of acoustic meati in the transversal plane with respect to the gravity line
Other: Static versus dynamic analysis — The use of clinical postural tests and instrumented movement analysis to evaluate the importance of muscle fatigue and compensation mechanisms
Other: Pre- versus postoperative analysis — The use of EOS stereo radiographic imaging and motion analysis to understand the compensation mechanisms in trunk, pelvis and lower limbs and the correlation between primary and secondary mechanisms.
  Arms: ASD with compensated sagittal misalignment; ASD with decompensated sagittal misalignment; ASD without sagittal misalignment
Other: Reliability of the dynamic evaluation — Repeated measurements of the different aspects of the dynamic evaluation protocol (strenght measurements of trunk muscles, balance evaluation and movement analysis) will serve to evaluate the test-retest reliability and intra-rater reliability of the different protocols

SUMMARY:
A good understanding of the principles of balance is vital to achieve optimal outcomes when treating spinal disorders. A complex interaction of the neuromotor system and muscular recruitment is necessary for ergonomic balance and deliberate displacement of the human body. Sagittal plane misalignment in spinal deformities challenges balance mechanisms used for maintenance of an upright posture. The occurrence of postoperative complications after spinal deformity correction like under-correction of sagittal misalignment, postoperative reciprocal changes in thoracic kyphosis, proximal junctional kyphosis and failure of instrumentation are possibly due to the current state-of-the art inadequate diagnostic work-up.

Investigators do not fully understand the roll of vision and exact strategy of recruitment of neuromuscular units (trunk, pelvis, lower limbs) in patients with sagittal plane misalignment during standing and walking. To understand this, a dynamic evaluation of individuals with spinal deformities is needed. Currently there is only very little research performed in the field of clinical balance tests and instrumented movement analysis in patients with spinal deformity.

The challenge for future studies is to further unravel the relation between trunk and lower limb movements, grouped into functional movement patterns. Moreover, additional information on trunk and lower limb kinetics and muscle activity (using dynamic electromyography (EMG)) will highly contribute to the understanding of this functional relationship, and will provide more in-depth insights into compensatory mechanisms of the trunk versus the lower limbs and vice versa.

DETAILED DESCRIPTION:
A good understanding of the principles of balance is vital to achieve optimal outcomes when treating spinal disorders. A complex interaction of the neuromotor system and muscular recruitment is necessary for ergonomic balance and deliberate displacement of the human body. Spinal alignment has to allow an individual to stand pain free with minimal muscular energy expenditure. This concept is reflected in the "Cone of Economy" principle by Jean Dubousset. Sagittal plane misalignment in spinal deformities challenges balance mechanisms used for maintenance of an upright posture. The current state of the art diagnostic work-up of spinal deformities is mainly a static 2D radiological evaluation in Scoliosis Research Society (SRS) free standing position with analysis of the spinopelvic parameters as described by Duval-Beaupmet and others.

Until now sagittal balance has been assessed by dropping a vertical plumb line from C7 vertebral body center and quantifying the distance of the sacral plate from this vertical (Sagittal Vertical Axis or SVA). Others measure the T1 spinopelvic inclination angle (T1-SPI). SVA, T1-SPI and pelvic tilt are correlated with self-reported disability and health related quality of life scores (HRQL) compared to age- and sex-related normal subjects.

Literature suggests a multifactorial etiology of impaired balance capacity with neurological or vestibular disease, muscular atrophy in mm erector spinae, increasing age, low back pain and history of spinal surgery. The occurrence of postoperative complications after spinal deformity correction like under-correction of sagittal misalignment, postoperative reciprocal changes in thoracic kyphosis, proximal junctional kyphosis and failure of instrumentation are possibly due to the current state-of-the art inadequate diagnostic work-up.

Investigators do not fully understand the roll of vision and exact strategy of recruitment of neuromuscular units (trunk, pelvis, lower limbs) in patients with sagittal plane misalignment during standing and walking. Several compensatory mechanisms in sagittal balance disorders are identified in the static situation. Intra-spinal mechanisms like hyperextension of lumbar discs, retrolisthesis of lumbar vertebrae, reduction of thoracic kyphosis, and pelvic back tilt and extra-spinal mechanisms like knee flessum and ankle extension are suggested to act as compensatory mechanisms. In literature, a strong correlation between the occurrence of knee flessum and lack of lumbar lordosis is seen. To understand these mechanisms a dynamic evaluation of individuals with spinal deformities is needed. Currently there is only very little research performed in the field of clinical balance tests and instrumented movement analysis in patients with spinal deformity. With regard to clinical balance tests the Fullerton Advanced Balance Scale (FAB scale) is presented as a reliable tool to predict wether or not higher-functioning older adults will fall. The FAB scale is a reliable and valid tool in Parkinson disease with minimal ceiling effect and shows promising results in detecting small balance disturbances.The use of these balance tests in patients suffering from spinal deformity with sagittal imbalance has not been validated in literature till now. Last but not least the use of instrumented movement analysis to examen gait in subjects with spinal deformity is unconventional. Subjects with fixed sagittal balance are reported to have a significant slower walking speed and poorer endurance score relative to age matched controls. An inadequate use of pelvic tilt during walking is also observed. Subjects with forward inclination of the trunk present with abnormal kinematics and kinetics of the lower limbs during walking compared to age- and sex-related normal subjects. When deformity exceeds the primary compensation mechanisms, additional mechanisms, such as crouch gait, are used to reorient the trunk to a more vertical position.

The currently used trunk model in movement analysis in UZ Leuven has been developed by Heyrman et al after the work of Leardini et al. Armand et al also considered the thorax not as one rigid segment and presented the use of an optimal marker placement set on the thorax for clinical gait analysis. However they did not include markers on the head. Heyrman et al showed in their study with cerebral palsy children (CP) that increased altered trunk movements during gait were related to a lower performance on the Trunk Control Measurement Scale (TCMS) in sitting, indicating the presence of an underlying trunk control deficit. These authors were thus able to show a correlation between a clinical postural test like the TCMS and trunk-and lower limb parameters during gait. However, they could not find a significant correlation between overall altered trunk movements and altered lower limb movements during gait in a CP population and concluded that observed thorax movements during gait, most likely are the resultant of both compensatory movements for lower limb deficits and an underlying trunk control deficit. The current concept of thinking is that in an adult spinal deformity population with sagittal plane misalignment the observed altered movements in the lower limbs during standing and gait are compensatory for the forward inclination of the trunk. The challenge for future studies is to further unravel the relation between trunk and lower limb movements, grouped into functional movement patterns. Moreover, additional information on trunk and lower limb kinetics and muscle activity (using dynamic electromyography (EMG)) will highly contribute to the understanding of this functional relationship, and will provide more in-depth insights into compensatory mechanisms of the trunk versus the lower limbs and vice versa.

ELIGIBILITY:
Inclusion Criteria:

* Pathological group

  1. Age >= 45 years
  2. Diagnosis of adult congenital, degenerative, idiopathic or iatrogenic spinal deformity
  3. Scoring at least 25 out of 30 on Mini Mental State Examination
  4. Ability to walk at least 50 meters distance independently without a walking aid
  5. Sagittal malalignment: PI-LL ≥ 25 degrees; sagittal vertical axis >5cm; pelvic tilt >25° and/or thoracic kyphosis > 60° and/or coronal malalignment: thoracic scoliosis 30 ≥ degrees; thoracolumbar/lumbar scoliosis ≥ 30 degrees; global coronal malalignment >3cm, posterior spinal fusion > 4 levels + iliac fixation.
  6. Ability and willingness of patient to attend follow-up visits and complete patient questionnaires
  7. Completed patient informed consent
* Control group

  1. Asymptomatic adults not suffering from a spinal deformity leading to a pathological sagittal alignment presenting as volunteer in the University Hospitals Leuven, Belgium
  2. Age >=45 years old
  3. Scoring at least 27 out of 30 on Mini Mental State Examination
  4. Ability to walk at least 1000 meters distance independently without a walking aid
  5. Ability and willingness of patient to attend follow-up visits and complete patient questionnaires
  6. Completed patient informed consent

Exclusion Criteria:

* Pathological group

  1. Age < 45 years old
  2. Absence of adult spinal deformity
  3. Scoring less than 25 out of 30 on Mini Mental State Examination
  4. Non-ability to walk at least 50 meters distance independently, with or without a walking aid.
  5. Missing patient informed consent
  6. Patients presenting with a neurological disease affecting balance other than Parkinson's disease such as stroke and/or Vestibular lesion
  7. Patients with a current history of diagnosed musculoskeletal disorders of the trunk and/or lower extremities affecting the motor performance such as severe hip arthrosis with or without flexion contracture, severe knee arthrosis, severe ankle arthrosis, severe leg length discrepancy (> 3 cm)
  8. BMI>30
* Control group

  1. Age < 45 years old
  2. Backpain and/or Sciatica at time of the study
  3. Presence of adult spinal deformity leading to a pathological sagittal alignment
  4. Scoring less than 27 out of 30 on Mini Mental State Examination
  5. Non-ability to walk at least 1000 meters distance independently without a walking aid
  6. Missing patient informed consent
  7. Patients presenting with a neurological disease affecting balance such as Stroke, Parkinson's disease and/or Vestibular lesion
  8. Patients with a current history of diagnosed musculoskeletal disorders of the trunk and/or lower extremities affecting the motor performance such as severe hip arthrosis with or without flexion contracture, severe knee arthrosis, severe ankle arthrosis, severe leg length discrepancy (> 3 cm)
  9. BMI > 27

Ages: 18 Years to 79 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 265 (Estimated)
Dates: Start 2016-01 (Actual); Primary Completion 2028-12 (Estimated); Study Completion 2028-12 (Estimated)

PRIMARY OUTCOMES:
Health-Related Quality of Life (HRQL) score | up to 2 years
  To evaluate the domains related to physical, mental, emotional, and social functioning
Postoperative state of the art radiographic evaluation (EOS/CT) | up to 2 years
  To investigate whether a state of the art correction of a spinal deformity causes a change in the dynamic function of the individual
Postoperative state of the art radiographic evaluation (EOS/CT) in correlation with HRQL | up to 2 years
  To investigate the correlation of radiographic evaluation with HRQL
3D motion analysis and balance tests | up to 2 years
  3D motion analysis and balance tests are combined to investigate the correlation with the static EOS stereo radiographic evaluation/CT/MRI
3D motion analysis and balance tests to investigate the dynamic function | up to 2 years
  3D motion analysis and balance tests are combined to investigate whether a state of the art correction of a spinal deformity causes a change in the dynamic function of the individual
3D motion analysis and balance tests in correlation with HRQL | up to 2 years
  3D motion analysis and balance tests are combined to investigate the correlation with HRQL (Health-Related Quality of Life)
Static EOS stereo radiographic evaluation | up to 2 years
  To investigate whether a state of the art correction of a spinal deformity causes a change in the dynamic function of the individual
Physical activity | up to 2 years
  Physical activity will be measured using a step counter (Garmin, Vivofit 4), which is a feasible and reliable parameter to measure physical activity in spinal surgery patients up to one-year post-op

SECONDARY OUTCOMES:
Falls Efficacy Scale-International (FES-I) | up to 2 years
  To measure the concerns about falling
EuroQol-5D-3L | up to 2 years
  To evaluate mobility, self-care, daily activities, pain / discomfort and anxiety / depression
Mini-Mental State Examination (MMSE) | up to 2 years
  To evaluate cognitive functions: attention and orientation, memory, registration, recollection, calculation, language and praxis.
Karnofsky Performance Score (KPS) | up to 2 years
  To determine the ability of patient to tolerate therapies in illness. The Karnofsky score runs from 100 to 0, where 100 is "perfect" health and 0 is death.
Cumulative Illness Rating Scale | up to 2 years
  To determine the presence of comorbidities. The scale format provides for 13 relatively independent areas grouped under body systems. Ratings are made on a 5-point "degree of severity" scale, ranging from "none" to "extremely severe".

CONTACTS AND LOCATIONS:
Overall Officials: Lieven Moke, Principal Investigator — Universitaire Ziekenhuizen KU Leuven
Locations (1):
- UZ Leuven, Leuven, Vlaams-Brabant, Belgium

IPD SHARING:
Plan to Share IPD: No